CLINICAL TRIAL: NCT06984198
Title: Assessing the Difference and Effectiveness of Art and Sand-play Therapy in Treating Post-traumatic Stress Disorders Among Syrian Refugee Children in Jordan
Brief Title: Comparing the Effectiveness of Art and Sand-play in Reducing PTSD Among Refugee Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Principal Investigator, khalid kheirallah, Professor of Epidemiology, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 464-2015
Record Dates: First submitted 2025-04-26; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: PTSD - Post Traumatic Stress Disorder
Keywords: Syrian refugee; PTSD; Sandplay; art therapy; mental health; Randomized trial; Children
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — Play Therapy; Art Therapy

STUDY DESIGN:
Intervention Model Description: Therapy Sessions In both the art and sand groups, each child will undergo 14 sessions, once per week. The first and last sessions will serve as pre and post-assessment sessions. The remainder 12 weeks will be the intervention period, where, depending on the child's randomized group assignment, they will either undergo no formal therapy (control), art, or sandplay therapy.
  SESSION 1: obtain the child's background history and consent, a pre-assessment of the child's condition using (HTQ).
  SESSION 2-13: Children in the sandplay and art therapy intervention groups will undergo their assigned therapies once a week.
  Session 14: HTQ, post intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sandplay therapy (Experimental): Sandplay Therapy - The objects involved in this form of therapy are: sandtray, sand, multiple figurines in all categories (people, animals, buildings, vehicles, vegetation, structures, natural objects and symbolic objects). The subject engaging in this therapy is instructed to build a sand picture with the minatures present. There is no time limit to these sessions; however, they tend to be 20-30 minutes long. Upon completion of their sand picture the child, if comfortable, may elaborate on their creation.
  Interventions: Behavioral: Sandplay Therapy
- Art therapy (Experimental): Art Therapy - The instruments used in this form of therapy are: a blank 8" x 11" paper and coloring utensils (markers, crayons, and color pencils). During each 30-minute session, the subject is informed to draw whatever they feel with the coloring utensils provided. Possible drawing topics may include: their family, a memory of their life back in their country of origin, or something from their imagination.
  Interventions: Behavioral: Art Therapy
- control (No Intervention): Standard care provided as per routine clinical practice.

INTERVENTIONS:
Behavioral: Sandplay Therapy — Sandplay Therapy - The objects involved in this form of therapy are: sandtray, sand, multiple figurines in all categories (people, animals, buildings, vehicles, vegetation, structures, natural objects and symbolic objects). The subject engaging in this therapy is instructed to build a sand picture with the minatures present. There is no time limit to these sessions; however, they tend to be 20-30 minutes long. Upon completion of their sand picture the child, if comfortable, may elaborate on their creation.
  Arms: Sandplay therapy
Behavioral: Art Therapy — Art Therapy - The instruments used in this form of therapy are: a blank 8" x 11" paper and coloring utensils (markers, crayons, and color pencils). During each 30-minute session, the subject is informed to draw whatever they feel with the coloring utensils provided. Possible drawing topics may include: their family, a memory of their life back in their country of origin, or something from their imagination.
  Other Names: art drawing
  Arms: Art therapy

SUMMARY:
Due to the political state of Syria, Jordan is experiencing a major increase in the number of Syrians seeking asylum each year, a quarter of which are children. The stressors these refugees are exposed to are described in three stages: (1) while in their country of origin; (2) during their escape to safety; and (3) when having to settle in a country of refuge.

The available literature shows consistently increased levels of psychological morbidity among refugee children, especially post-traumatic stress disorder (PTSD). It is argued that mental health clinics could use creative art therapies as a means of reaching out to war refugees in their communities who may not respond to traditional therapy. The difference in effectiveness between art and sand-play therapy, two models of nonverbal psychosocial therapy, on Syrian refugee children with PTSD, will be evaluated using a pretest-posttest control group design with 90 preadolescents (ages 6-12) exhibiting PTSD. Children will be randomized into two experimental groups (n = 30 for each) to receive sandplay or art therapy for 12 weeks, while the control group (n = 30) will receive no formal treatment. The effectiveness of each form of therapy will be determined using a questionnaire and then compared within and between group(s). Further statistical analysis will be used to determine which therapy was more effective in mitigating PTSD.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) involves severe symptoms like re-experiencing trauma, avoidance, and hyperarousal, lasting more than a month and causing significant distress or functional impairment. Common treatments include EMDR and TF-CBT, but over 30% of patients do not benefit, especially those with complex trauma or poor verbal memory. Sand-play therapy is a nonverbal psychotherapeutic technique where clients create a "sand-world" using miniatures in a sandbox. Developed by Margaret Lowenfeld and later expanded by Dora Kalff, it offers therapeutic value through its multidimensional nature, narrative potential, access to preverbal memories, and accessibility without requiring special skills. It allows individuals to express internal experiences symbolically, supporting emotional healing in a safe, non-judgmental environment. Sand-play therapy uses a sand-tray and miniature objects like people, animals, buildings, and natural elements to help children express their inner experiences nonverbally. The process typically has two stages. First, the child creates a "sand-world" in silence, without any input from the therapist, allowing for personal, unconscious expression. Therapists avoid interpretations at this stage, respecting that each object can have unique meaning to the child.

In the second stage, the child may choose to explain the story behind their creation, helping them clarify emotions and gain insight. This encourages the release of negative feelings and memories stored in the unconscious. While some therapists interpret symbols based on the child's background, interpretation remains debated. Many believe that imposing meaning is unnecessary, as healing can occur naturally through the child's self-expression.

Furthermore, while counselors practicing from a Jungian perspective commonly use interpretation of children's pictures as a component of the therapeutic process, others argue that interpretation is not only unnecessary but also inappropriate. It is suggested that symbols are arbitrary and have unique meanings for individuals and, as such, their subjective nature must be respected. It is also noted that because sand-play allows issues to be resolved on an unconscious level, interpretation is seldom needed. Thus, for the purposes of this research we refrain from analyzing and interpreting the children's sandboxes to devote the counseling sessions just to the therapeutic value of sand-play therapy.

Overall, the counselor's primary role is to provide a safe and emotionally permissive environment for the child's expression of feelings and experiences. The child should be encouraged to express whatever he or she is experiencing with the freedom to determine how materials are used and what scenes are created in the sand. Hence, sand-play therapy can be considered as a form of play therapy and its basis in play is one factor that makes it particularly worthy of consideration for use in school contexts. It is suggested that this innate inner healing mechanism can reveal those things that need to be remembered, felt, released, or integrated and, as such, children are viewed as being capable of actively directing the resolution of their own concerns.

It is known that play is the singular central activity of childhood and is a spontaneous, enjoyable, voluntary and non-goal directed activity. It gives concrete form and expression to children's inner worlds and provides them with a symbolic language for self-expression, which is what is experienced when the child undergoes sand-play therapy. It has been suggested that in a counseling context, play is to the child, what verbalization is to the adult and literature pertaining to the use of therapeutic play with children frequently describes play as their language and toys as their words. It is known that in traditional counseling approaches, when children experience enormously complex feelings and thoughts in relation to the events in their lives, they often have difficulty trying to communicate these verbally in the counseling context. Using therapeutic techniques that are based in play provides the most natural and non-threatening means for children to communicate and act out sensitive material related to frightening and difficult situations.

In sand-play therapy, interpretation of a child's creation is a debated practice. While some Jungian therapists view it as helpful, others argue that symbols are personal and subjective, making formal interpretation unnecessary and potentially inappropriate. Since healing often occurs unconsciously, interpretation is rarely needed. Therefore, this study focuses solely on the therapeutic value of the child's self-expression without analysis or interpretation.

The therapist's role is to create a safe, supportive space where children feel free to express emotions and experiences through play. Sand-play is considered a form of play therapy, which aligns with how children naturally communicate-using play as their language and materials as their words. Play is spontaneous and non-goal-oriented, allowing children to safely explore and express complex feelings that may be difficult to verbalize. This makes play-based therapy especially effective for helping children process trauma and other emotional challenges in a natural, non-threatening way.

Much like sand-play therapy, art therapy is also a form of play therapy where the client engages in a nonverbal expression. Characteristic for art therapy is the methodical use of means as drawing, painting, collage, and sculpting to shape and express feelings, thoughts and memories. Art therapy is a distinguished form of treatment by active performance and experience with art materials, by visual and concrete character of the process, as well as by the result of art making. In clinical practice, the aim of art therapy is to elicit processes of change, development, and acceptance, using art in a purposeful and methodical way in the treatment of psychosocial problems and mental disorders. Experts have discussed the benefits of art therapy in the treatment of PTSD in adults, where decreases in primary PTSD symptoms have been reported as outcomes of art therapy.

Although there are no previously published reports of sand-play therapy for individuals with PTSD as a result of war trauma, a brief literature review yielded several studies of sand-play work with other special populations. Sand-play therapy has successfully been used with a range of disorders and a variety of situations among children and adults, including adjustment disorders, affective disorders, eating disorders, and abuse. Studies specific to children who have experienced abuse reported more chaotic, disorganized sand-play productions, fewer nature scenes, fewer objects, and reduced conflict resolution compared to control groups. Thus, the primary significance of this study will be that it will further contribute to the clinical uses of sandplay and art therapy. More importantly, it will provide evidence to the merits of sand-play therapy for war refugees with PTSD. For instance, it can be difficult to reach refugee populations within a community whose culture and language are different from the majority, but finding other means of communicating can make a real difference for these individuals as they find safety and understanding by working on and sharing special creative projects. Thus, these forms of therapy can serve a greater advantage to these communities.

Art therapy, like sand-play, is a form of nonverbal play therapy that uses creative activities such as drawing, painting, and sculpting to help individuals express emotions, thoughts, and memories. It encourages personal growth and healing through the creative process and has been shown to reduce PTSD symptoms in adults.

Although no studies have yet explored sand-play therapy for war-related PTSD, it has been successfully used with other groups, including children with adjustment disorders, abuse trauma, and emotional difficulties. Children who have experienced abuse often create more disorganized scenes with fewer positive elements compared to others.

This study aims to expand the use of sand-play and art therapy by testing their effectiveness in treating PTSD among Syrian refugee children in Jordan. These therapies offer a culturally sensitive, nonverbal way to reach children who may struggle with traditional talk-based methods, helping them process trauma through creativity and self-expression.

Goal and Objective: To determine the difference in effectiveness between art and sandplay therapy, as compared to each other and to the control group, on Syrian refugee children with PTSD living in Jordan.

Subject Exclusion and Inclusion Criteria:

Syrian children, ages 6-12 that are refugees living in Jordan as a result of the Syrian Civil War, will be considered for this study. To be included in the current study, children should also experience trauma related to the war as diagnosed by the treating physician. Participating children should not have pre-existing psychosocial issues.

Randomization:

Children (N=90) will be randomized into three groups (n=30 for each): Sand, Art, and Control groups. An even distribution of ages and gender will be maintained in this process.

Assessment (Instruments):

Harvard Trauma Questionnaire checklist will be used to assess the mental health status of children in a pre and post intervention format. The checklist inquiries about a variety of trauma events, as well as the emotional symptoms considered to be uniquely associated with trauma. The scoring method used in this study will be adapted from this questionnaire and will include questions to help determine the children's PTSD severity, which will be split into three degrees: mild, moderate, and severe. The questionnaire comprises of 16 questions, each with a rating of 1-4. Subjects with scores between 16-32, 33-48, or 49-64 were considered mild, moderate, or severe, respectively. HTQ checklist will be translated into Arabic, and then back translated to ensure validity and reliability.

Sand-play Therapy - The objects involved in this form of therapy are: sand-tray, sand, multiple figurines in all categories. The subject engaging in this therapy is instructed to build a sand picture with the miniatures present. There is no time limit to these sessions; however, they tend to be 20-30 minutes long. Upon completion of their sand picture the child, if comfortable, may elaborate on their creation.

Art Therapy - The instruments used in this form of therapy are: a blank 8" x 11" paper and coloring utensils. During each 30-minute session, the subject is informed to draw whatever they feel with the coloring utensils provided. Possible drawing topics may include: their family, a memory of their life back in their country of origin, or something from their imagination.

Therapy Sessions:

In both the art and sand groups, each child will undergo 14 sessions, once per week, for duration of 14 weeks. The first and last sessions will serve as pre and post-assessment sessions, respectively. The remainder twelve weeks will be the intervention period, where, depending on the child's randomized group assignment, they will either undergo no formal therapy, art, or sand-play therapy.

SESSION ONE: Establish a safe environment for the child, obtain the child's background history and consent for participation in the study, and take a pre-assessment of the child's condition to determine the severity of their PTSD as established by their answers provided on their translated Harvard Trauma Questionnaire.

SESSION 2-13: Children in the sand-play and art therapy intervention groups will undergo their assigned therapies once a week. The therapist present during each session will follow the guidelines outlined in the manual of each form of therapy. Expected duration of each session is one hour where 15 minutes will serve as an opportunity to engage in an optional verbal explanation of their creation. The children will be given the option to not participate in each week's session. Each child's sand-tray or art pieces will be photographed for documentation and analysis purposes.

SESSION 14: The last session will serve as a closing meeting for their involvement in the study. Post-assessment will also be taken using the same questionnaire used at the beginning of the study.

Data Analysis:

Mean score of HTQ checklist will be calculated pre and post intervention for both experimental groups and the control group. In each group, the mean change over the 12-week intervention will be calculated and compared with the control group and the other therapy group. Paired t-test will be used to compare the pre-post mean in each group. T-test will be used to compare the mean difference between each group and the control and between the two therapy groups. A P-value of 0.05 will be used to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Syrian refugee children living in Jordan as a result of the war/conflict in Syria,
* Ages between 6 and 12 years at the time of the study.
* Reported to have experienced trauma related to the war/conflict in Syria (e.g. witnessed death, shrapnel injuries, and/or any forms of war violence) as diagnosed by the treating physician.
* Lack of any pre-existing psychosocial issues.
* Ability to secure parent or guardian consent.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
HTQ | Week 1, pre-intervention, and then week 14, post-intervention.
  HTQ: Harvard Trauma Questionnaire, translated into Arabic. Harvard Trauma Questionnaire (HTQ) checklist will be used to assess the mental health status of children in a pre and post intervention format. The checklist, written by Harvard Program in Refugee Trauma (HPRT), inquires about a variety of trauma events, as well as the emotional symptoms considered to be uniquely associated with trauma (Harvard Trauma Questionnaire, 2011). The scoring method used in this study will be adapted from this questionnaire and will include questions to help determine the children's PTSD severity, which will be split into three degrees: mild, moderate, and severe. The questionnaire used (please refer to Appendix B for a detailed outline of the instrument) comprises of 16 questions, each with a rating of 1-4 (1: not at all and 4: extremely). Subjects with scores between 16-32, 33-48, or 49-64 were considered mild, moderate, or severe, respectively. HTQ checklist will be translated into Arabic.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Alzoubi, MD, PhD, Principal Investigator — Medical School of Jordan University of Science and Technology; Khalid A Kheirallah, PhD, Study Director — Medical School of Jordan University of Science and Technology
Locations (1):
- Zad Children Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
IPD were not actually collected as there was only age and sex of the participant along with their drawings that were needed as part of the data collection. This will be shared for reasonable use if needed as per the IRB requirements.
Supporting Information: Study Protocol
Time Frame: Dec 2025

REFERENCES:
- [Background] Lee HJ, Na K, Kwon MS, Kim H, Kim KS, Paik YK. Quantitative analysis of phosphopeptides in search of the disease biomarker from the hepatocellular carcinoma specimen. Proteomics. 2009 Jun;9(12):3395-408. doi: 10.1002/pmic.200800943. PMID 19562805
- [Background] Jones JM, Jolly RD. Dwarfism in Hereford cattle: a genetic morphological and biochemical study. N Z Vet J. 1982 Dec;30(12):185-9. doi: 10.1080/00480169.1982.34937. PMID 16030843
- [Background] Garcia Vallejo R, Martinez Hernandez E, Amal Selfa R, Canada DA. [Working with the scientific method]. Rev Enferm. 2004 Jan;27(1):15-8. Spanish. PMID 15040591
- [Background] Goggs R, Boag AK, Chan DL. Concurrent immune-mediated haemolytic anaemia and severe thrombocytopenia in 21 dogs. Vet Rec. 2008 Sep 13;163(11):323-7. doi: 10.1136/vr.163.11.323. PMID 18791206
- [Background] Low N, Cowan F. Genital chlamydial infection. Clin Evid. 2002 Dec;(8):1601-7. No abstract available. PMID 12603957
- [Background] Ng MH, Choo YM, Ma AN, Chuah CH, Hashim MA. Separation of vitamin E (tocopherol, tocotrienol, and tocomonoenol) in palm oil. Lipids. 2004 Oct;39(10):1031-5. doi: 10.1007/s11745-004-1327-y. PMID 15691027
- [Background] Larsen FS. Is it worthwhile to use cerebral microdialysis in patients with acute liver failure? Neurocrit Care. 2006;5(3):173-5. doi: 10.1385/NCC:5:3:173. No abstract available. PMID 17290083
- [Background] Carmichael, Karla Delle. "Sand Play as an Elementary School Strategy." Elementary School Guidance & Counseling, vol. 28, no. 4, 1994, pp. 302-07. JSTOR, http://www.jstor.org/stable/42871132.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: 6. Statistical Analysis Plan (2014-04-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT06984198/Prot_SAP_000.pdf